CLINICAL TRIAL: NCT03228212
Title: Evaluation of Approved and Investigational Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5960
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Results first posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL/CONTROL (Experimental): Enrolled subjects will be habitual wearers of spherical contact lenses between the ages of 18 and 49 years old. Subjects will wear the Test and Control contact lenses bilaterally for approximately 2 weeks each on a daily wear basis. Subjects will be randomly assigned to one of the two lens wear sequences, (TEST/CONTROL/CONTROL)
  Interventions: Device: CONTROL; Device: TEST
- CONTROL/TEST/TEST (Experimental): Enrolled subjects will be habitual wearers of spherical contact lenses between the ages of 18 and 49 years old. Subjects will wear the Test and Control contact lenses bilaterally for approximately 2 weeks each on a daily wear basis. Subjects will be randomly assigned to one of the two lens wear sequences, (CONTROL/TEST/TEST)
  Interventions: Device: CONTROL; Device: TEST

INTERVENTIONS:
Device: CONTROL — ACUVUE OASYS
Device: TEST — senofilcon A with new UV blocker

SUMMARY:
This study is a randomized, 5-visit, partial subject masked, 2x3 bilateral crossover, dispensing clinical trial. During the study, each test article will be worn in a daily wear modality for at least 6 hours per day and 5 days per week for approximately 2 weeks each. The subject will wear either the Test or Control article twice and the other study article once. The primary objective of this study is to demonstrate that the Test lens works as well, if not better compared to the Control lens with respect to CLUE (Contact Lens User Experience) comfort, Slit Lamp findings, and Distance Monocular logMAR Visual Acuity. This study will also aim to show acceptable lens fit for subjects wearing the Test lens.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following inclusion criteria to be enrolled in the study:

  1. The subject must read and sign the Informed Consent form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Healthy adult males or females age ≥18 and ≤49 years of age with signed informed consent. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them.
  4. The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and - 6.00 Diopter (D).
  5. The subject's refractive cylinder must be ≤ 1.00D in each eye.
  6. The subject must have visual acuity best correctable to 20/25+3 or better for each eye.
  7. Subjects must own a wearable pair of spectacles.
  8. The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of Daily Wear per day, at least 5 days per week, for a minimum of 1 month prior to the study) and willing to wear the study lenses on a similar basis.
  9. Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week
  10. The subject must have normal eyes (i.e., no ocular medications or infections of any type).

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
  2. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
  3. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral (e.g., Chlor-Trimeton, and Benadryl) and ophthalmic antihistamines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), oral and ophthalmic Beta-adrenergic blockers (e.g., Propranolol, Timolol, and Practolol), systemic steroids, and any prescribed or over the counter (OTC) ocular medication.
  4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion.
  5. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), LASIK, etc.).
  6. Any Grade 3 or greater slit lamp findings (e.g.., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
  7. Any known hypersensitivity or allergic reaction to Optifree®PureMoist® multi-purpose care solution or Eye-Cept® rewetting drop solution
  8. Any ocular infection, allergy or clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca, ocular hypertension), or ocular conditions (e.g. strabismus), which might interfere with the study.
  9. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
  10. Toric, extended wear, monovision or multi-focal contact lens correction.
  11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  12. Participation in clinical trials involving the Test lens within 3 months prior to study enrollment.
  13. History of binocular vision abnormality or strabismus.
  14. Employee, relative or friends of employees of any ophthalmic company, or investigational clinic (e.g., Investigator, Coordinator, Technician).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Dr. James Weber & Associates, PA, Jacksonville, Florida
  - Vue Optical Boutique, Jacksonville, Florida
  - VisionCare Associates, East Lansing, Michigan
  - Pickens Family Eye Care, Pickens, South Carolina
  - William J. Bogus, OD, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 133 subjects were enrolled into this study. Of the enrolled subjects, 130 were dispensed at least one study lens and 3 subjects failed to meet all eligibility criteria. Of the dispensed subjects 127 completed the study while 3 subjects were discontinued.
Groups:
- Test/Control/Control: Subjects that wore the Test lens during the first period, and the control lens during the second and third period of the study.
- Control/Test/Test: Subjects that wore the Control lens during the first period and the Test lens during the second and third period.
Period: Period 1
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 65 | 65
Completed | 64 | 64
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — no longer meets eligibility criteria | 0 | 1
Period: Period 2
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 64 | 64
Completed | 63 | 64
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Period 3
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 63 | 64
Completed | 63 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dispensed Subjects: All subjects that were dispensed at least one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.6 (7.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  American Indian or Alaska Native | 2
  Black or African American | 12
  White | 111
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average comfort score from the 3 study periods was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Test: Subjects that wore the Test lens during any of the 3 periods of the study.
- Control: Subjects that wore the Control lens during any of the 3 periods of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 121 | 121
Units on a Scale | 67.509 (23.8724) | 61.185 (24.2024)
Statistical Analysis 1: Comparison: Test vs Control; It was calculated that 60 participants randomized in a 1:1 fashion between the two sequences would have at least 80% power to detect a 5 points difference in mean overall comfort at the 2-week follow-up. Sample size was determined using Stroup's Method (alpha=0.05); Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE scores; Bayesian multivariate normal random-effe; A 95% Credible Interval for the Posterior mean difference between the Test and Control was used to test for non-inferiority; Mean Difference (Final Values) = 5.1, 95% CI 2-sided [1.16 to 9.09], Standard Deviation 2.0 — Mean difference was calculated as Test - Control

2. Primary Outcome: Distance Monocular LogMAR Visual Acuity
Description: Distance Monocular LogMAR visual acuity was assessed at 4 meters using an ETDRS chart at the 2-week follow-up for each subject eye during each of the three study periods. The average visual acuity for each lens type from the 3 study periods was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 65 | 65
Number analyzed (Eyes) | 130 | 130
logMAR | -0.095 (0.0831) | -0.075 (0.0806)
Statistical Analysis 1: Comparison: Test vs Control; It was calculated that 40 participants randomized in a 1:1 fashion between the two sequences would have at least 80% power to detect a 0.05 difference in LogMAR visual acuity at the 2-week follow-up. Sample size was determined using simulations methods for repeated measures; Test type: Non-Inferiority — A non-inferiority margin of 0.05 logmar was used. This margin corresponds to a half line difference; Bayesian multivariate normal random-effe; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [0.01 to 0.03], Standard Deviation 0.00621 — Mean difference was calculated as Test - Control

3. Primary Outcome: Contact Lens Fitting Acceptance Rate
Description: Contact lens fitting acceptance was assessed for each subject eye using a biomicroscope at post lens insertion and the 2-week follow-up. Lens fit was a binary variable where acceptable lens fit=1 and unacceptable lens fit=0. The proportion of eyes with acceptable lens fit was reported for each lens. The lens fit acceptance rate for both post lens fitting at the 2-week follow-up was reported for each lens type.
Time Frame: Up to 2-Week Follow-up
Population: Subjects that completed all study visits.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 65 | 65
Number analyzed (eyes) | 130 | 130
proportion of eyes | 1 | 1
Statistical Analysis 1: Comparison: Test; It was calculated that 70 participants randomized in a 1:1 fashion between the two sequences would have at least 80% power to detect a the 2-week follow-up. Sample size was determined using simulations methods for repeated measures. Analysis was only performed on eyes wearing the Tesl lens; Test type: Non-Inferiority — A non-inferiority margin of 90% was used. Lower limit of 95% credible interval was compared to 90%; Bayesian Methods; Bayesian Methods-Jefferys prior for binomial proportion was used to calculate 95% credible interval; proportion = 0.992, 95% CI 2-sided [0.96 to 1]

4. Primary Outcome: Number of Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). This was performed on each subject eye at every study visit (baseline, unscheduled visits and 2-week follow-up). The data was then dichotomized into two groups. Those with grade 3 or higher and those with grade 2 or lower. The number of SLF with grade 3 or higher by lens was reported.
Time Frame: Up to 2-Week Follow-up
Population: Subjects that were dispensed at least one study lens.
Measure: Number; unit: Slit Lamp Finding
Units Other Than Participants: Eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 65 | 65
Number analyzed (Eyes) | 130 | 130
Slit Lamp Finding | 0 | 1
Statistical Analysis 1: Comparison: Test vs Control; It was calculated that 120 participants randomized in a 1:1 fashion between the two sequences would have at least 80% power to detect 5% difference between the Test and Control lens with respect to the proportion of eyes with Grade 3 or higher slit lamp findings across all study visits. Sample size was determined using simulations methods. Sample size for this study was primarily driven by the slit lamp findings; Test type: Non-Inferiority — A non-inferiority margin of 5% was used. Upper limit of the 95% credible interval was compared to 5%; Bayesian beta-binomial model; Bayesian beta-binomial model for correlated binary data; Mean Difference (Final Values) = -0.0043, 95% CI 2-sided [-0.0237 to 0.0129], Standard Deviation 0.0089 — Mean difference calculated as Test - Control

5. Secondary Outcome: Overall Quality of Vision
Description: Overall quality of vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average vision score from the 3 study periods was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test | Control
Number analyzed (Participants) | 121 | 121
Units on a Scale | 69.16 (20.362) | 60.329 (22.289)
Statistical Analysis 1: Comparison: Test vs Control; Sample size calculations were based on the primary endpoints; Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE scores; Bayesian multivariate normal random-effe; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.2, 95% CI 2-sided [3.69 to 10.74], Standard Deviation 1.8 — Mean difference was calculated as Test - Control

6. Secondary Outcome: Overall Handling
Description: Overall Handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average handling score from the 3 study periods was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test | Control
Number analyzed (Participants) | 121 | 121
Units on a Scale | 72.11 (20.046) | 66.79 (20.007)
Statistical Analysis 1: Comparison: Test vs Control; Sample size calculations were based on the primary endpoints; Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE scores; Bayesian multivariate normal random-effe; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [0.36 to 6.29], Standard Deviation 1.5 — Mean difference was calculated as Test - Control

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 6 weeks per subject.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/130
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/130
Other Adverse Events (participants affected / at risk) | 0/130 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT03228212/Prot_SAP_000.pdf